CLINICAL TRIAL: NCT03983928
Title: A Phase Ib, Open-label, Single Center, Non-randomized Study for Safety and Efficacy of TQB2450 Combined With Anlotinib in Subjects With Advanced Mutation Positive Non-Small Cell Lung Cancer
Brief Title: Study of TQB2450 Combined With Anlotinib in the Treatment of Mutation Positive Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ib-11
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 Combined with Anlotinib (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450; Drug: Anlotinib

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
Drug: Anlotinib — a multi-target receptor tyrosine kinase inhibitor

SUMMARY:
This is an open-label, single center, non-randomized, phase Ib trial to evaluate safety and efficacy of TQB2450 injection combined with anlotinib in patients with advanced mutation positive non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Understood and signed an informed consent form.
2. 18 years and older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, life expectancy≥ 12 weeks.
4. Histologically or cytologically confirmed mutation positive non-small cell lung cancer according to 8th International Association for the Study of Lung Cancer (IASLC) edition.
5. Has measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
6. Adequate organ system function, defined as follows:

   1. absolute neutrophil count (ANC) ≥ 1.5×10^9/L, platelets (PLT) ≥ 100×10^9/L, hemoglobin (Hb)≥ 90g /L;
   2. total bilirubin (TBIL) ≤ 1.5×ULN；alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN (without liver metastasis) or ≤ 5.0 × ULN (with liver metastasis), Creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 ml/min;
   3. Urine protein < ++，or urine protein ≥ ++ concomitant with content of 24-hour urinary protein <1.0 g;
   4. international normalized ratio (INR) ≤ 1.5×ULN, activated partial thromboplastin time (APTT) ≤ 1.5×ULN;
   5. left ventricular ejection fraction (LVEF) ≥ 50%;
7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ; No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

Exclusion Criteria:

1. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization except of cured in situ carcinoma of the cervix, non-melanoma skin cancer and superficial bladder carcinoma.
2. Has severe hypersensitivity reactions after taking other monoclonal antibodies.
3. Has hypersensitivity reactions after taking anlotinib.
4. Has prior therapy with anlotinib, anti-programmed cell death (PD)-1, anti-PD-L1 or other immunotherapy against PD-1/PD-L1.
5. Has any active autoimmune disease or history of autoimmune disease, such as autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis, asthma patients who need bronchiectasis for medical intervention; Subjects with the vitiligo without systemic treatment, psoriasis, alopecia, well-controlled type I diabetes mellitus, hypothyroidism stable on hormone replacement will not be excluded from this study.
6. Has multiple factors affecting oral medication, such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.
7. Has clinical significance of thyroid dysfunctions within 6 months prior to enrollment, and even though medical therapy, thyroid function can not return to normal or no clinical significance.
8. Has central nervous system (CNS) metastases without local therapy of lesion.
9. Radiograph (within 28 days before enrollment) showed that the tumor surrounded important blood vessels, and the investigators determined that entering the study would cause bleeding risk.
10. Hemoptysis (defined as coughing out or spitting out ≥ 1 teaspoon of blood or small blood clots or hemoptysis without sputum) within 28 days before enrollment , not including bloody sputum.
11. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration.
12. Has any of the following severe acute complications:

    1. Unstable angina and/or congestive heart failure or vascular disease requiring hospitalization within 12 months, or other cardiac impairments determined by the investigator, which may affect the evaluation of drug safety; Myocardial infarction or ischemia with ST elevation ≥ 2 mm indicated by electrocardiogram (ECG);
    2. Has pulmonary infections and/or acute bacterial or fungal infections requiring intravenous antibiotic therapy;
    3. Has clinical jaundice caused by liver dysfunction;
13. Virological test indicates one of the following items before enrollment:

    1. HBsAg positive and HBV DNA ≥ 1 × 10^3 copies/mL;
    2. Anti-HCV positive and HCV virus titer detection value exceeds the upper limit of normal value;
    3. HIV positive;
14. Has participation in an anti-tumor clinical trial within 28 days prior to the first administration.
15. Has serious affecting safety or treatment compliance concomitant diseases, according to the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate （ORR） | up to approximately 12 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to approximately 12 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to approximately 15 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Disease control rate（DCR） | up to approximately 12 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China